CLINICAL TRIAL: NCT01587729
Title: IMI PROTECT (Work Package 2): Use of Antidepressants and Risk of Hip and/or Hip/Femur Fracture
Brief Title: IMI PROTECT(WP2): Antidepressants & Fractures
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115734; WEUKBRE5556 (Other: GSK)
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Depression, Postpartum
Keywords: Hip/femur fracture; antidepressants
MeSH Terms: conditions — Depression, Postpartum | interventions — Selective Serotonin Reuptake Inhibitors; Antidepressive Agents

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with a diagnosis of hip or femur fracture: All patients of the study population with a record/diagnosis of a first fracture of the hip or femur during the study period regardless of whether they have a history of past fractures. When the patient has a history of hip or hip/femur fracture, a minimum of 12 months should have elapsed between the two episodes for a current fracture to be considered a new event.
  Interventions: Drug: Tricyclic AD (TCAs) and selective serotonin re-uptake inhibitors (SSRIs) antidepressants
- Patients without a diagnosis of hip or femur fracture: All patients of the study population without a record/diagnosis of a fracture of the hip or femur during the study period
  Interventions: Drug: Tricyclic AD (TCAs) and selective serotonin re-uptake inhibitors (SSRIs) antidepressants

INTERVENTIONS:
Drug: Tricyclic AD (TCAs) and selective serotonin re-uptake inhibitors (SSRIs) antidepressants — TCA or SSRI prescription during the study period between January 1, 2001 and December 31, 2009. The TCAs and SSRIs administered to the patients include paroxetine and escitaloprim.

SUMMARY:
The studies described in this protocol are all performed within the framework of PROTECT (Pharmacoepidemiological Research on Outcomes of Therapeutics by a European ConsorTium) Workpackage 2 and Workgroup 1. Primary aim of these studies is to develop, test and disseminate methodological standards for the design, conduct and analysis of Pharmacoepidemiological (PE) studies applicable to different safety issues and using different data sources. To achieve this, results from PE studies on five key adverse events (AEs) performed in different databases will be evaluated. Therefore, emphasis will be on the methodological aspects of the studies in this protocol and not on the clinical consequences of the association under investigation.

Fracture of the proximal end of the femur or hip is associated with considerable morbidity and mortality. Hip/femur fractures impair quality of life and impose a considerable economic burden, and occur with 20% mortality rate within the first year. Antidepressants (AD), mainly tricyclic AD (TCAs) and selective serotonin re-uptake inhibitors (SSRIs) have been associated with fractures in several studies. A review of 13 observational studies showed risk ratios ranging from 1.2 to 3.7 for current TCA users and a wide range of 1.5 to 8.6 for SSRI users. The majority of the studies in the aforementioned review reported increased risks of fractures in general with SSRIs use and more mixed risk outcomes for TCA use. Several mechanisms underlying this adverse effect have been postulated in the literature: e.g. through decrease in bone mineral density (BMD) or through blocking the serotonin transporter activity (5-hydroxytryptamine re-uptake) and hence affecting bone metabolism and structure or simply by falling or through co-morbidities such as depression itself. Previous observational studies differ in design, conduct and analysis of the considered association with varying degree of accounting for confounders. Confounding factors such as depression and other co-morbidities, previous fractures, concomitant drug use and lifestyle factors such as smoking have usually not been accounted for in most of the studies. In addition, small sample size, different methods used to ascertain exposure, selection bias and lack of data on compliance as well as important covariates limit the use of these results in benefit-risk analyses. Furthermore, studies evaluating different types of SSRI and TCA are few and dose-response relationship for most of the AD remains to be studied. We will study effects of cumulative exposure focusing on acute (less than 6 months) and long term exposure (at least 5 years) and doses of exposure.

The objective of the study is to assess the association between AD use and hip/femur fracture using different study designs (descriptive, cohort, nested case-control and case crossover) across different databases and to compare the results between and across databases and designs. This is to evaluate the impact of design/database /population difference in the outcome of the studies association.

Data will be collected from the following databases: The Health Improvement Network [(THIN]), a UK-based primary care electronic medical record database, the Dutch Mondriaan project (a primarily general physician based database with some linkage to survey data from the Netherlands), Base de Datos para la Investigación Farmacoepidemiológica en Atencion Primaria [(BIFAP] (Spanish primary care database)), and the Bavarian statutory health insurance physicians' association database (German health insurance database from primary and secondary care).

ELIGIBILITY:
For the descriptive study:

Inclusion Criteria:

* patients who have at least one year of enrolment with the GP
* patients who are at least 18 years of age
* patients who have at least one antidepressant prescription

Exclusion Criteria:

* patients with an antidepressant prescription within 6 months prior to study start
* patients missing information on sex and age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all patients included in the period of valid data collection for each of the databases. The study period will be defined from January 1, 2001 to December 31, 2009. Information on the use of antidepressants and occurrence of hip/femur fracture will be obtained from individual databases comprising of medical records of general practitioners and/or claims data where prescription and diagnosis data are recorded.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
First fracture of hip or femur during the study period | Up to nine years following drug exposure
  Fracture will be defined using International Classification of Diseases version 10 (ICD-10) codes in the Bavarian database, READ codes in THIN and International Classification of Primary Care (ICPC-2) in BIFAP and Mondrian

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline